CLINICAL TRIAL: NCT02668978
Title: Prospective Randomized Clinical Trial to Prevent Air Leaks After Lung Resection With Hemopatch™ Sealing Hemostat: SEALLS (Sealing Evaluation of Air Leaks After Lung Surgery) Trial
Brief Title: SEALLS (Sealing Evaluation of Air Leaks After Lung Surgery) Trial Using HEMOPATCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Quirón Madrid University Hospital (Other)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Principal Investigator, Javier MORADIELLOS, Associate Chief of Thoracic Surgery, Quirón Madrid University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEALLS
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: LUNG DISEASES
Keywords: lung surgery; air leak; prevention
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopatch™ (Experimental): Hemopatch™ sealing hemostat
  Interventions: Device: Hemopatch™ Sealing Hemostat
- Control (Active Comparator): Standard surgical technique
  Interventions: Procedure: Standard surgical technique

INTERVENTIONS:
Device: Hemopatch™ Sealing Hemostat — Hemopatch™ application over lung resection areas
  Arms: Hemopatch™
Procedure: Standard surgical technique — Lung resuturing or restapling
  Arms: Control

SUMMARY:
The primary objective is to assess the efficacy and safety of HEMOPATCH™ Sealing Hemostat in reducing the incidence and duration of air leaks after lung resection compared to standard techniques.

Hypothesis: "The routine application of HEMOPATCH Sealing Hemostat on the visceral pleura in lung resection areas, during lung resection procedures, is more EFFICIENT to reduce the incidence and duration of prolonged air leaks as compared to standard surgical measures."

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years who are able to give their informed consent
* Patients undergoing lung resection surgery for either malignant or benign conditions including:

  * Lobar and sublobar resections
  * Open, video-assisted thoracoscopic or robotic surgeries
  * Diagnostic or therapeutic procedures

Exclusion Criteria:

* Traumatic pulmonary contusion or laceration
* Lung reduction surgery
* Planned removal of more than 10 lung lesions
* Pneumonectomy
* Known hypersensitivity to bovine protein
* Known hypersensitivity to Brilliant Blue FCF (E133)
* Presence of active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative air leaks | Within first 30 postoperative days
  Duration of postoperative lung air leaks expressed in hours

CONTACTS AND LOCATIONS:
Locations (1):
- Quirónsalud Madrid University Hospital, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No